CLINICAL TRIAL: NCT04381481
Title: Studying the Impact of Product Packaging in a Virtual Store Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-3227; K01HL147713 (NIH)
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Control beverage, text snack (Experimental): The participant will see fruit drinks with no nutrition claims (task 1). They will see a snack with a text warning "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Control Drink: No nutrition claim; Behavioral: Experimental snack: Text warning
- Control beverage, control snack (Experimental): The participant will see fruit drinks with no nutrition claims (task 1). They will see a snack with a barcode label (control label) (task 2).
  Interventions: Behavioral: Control Drink: No nutrition claim; Behavioral: Control snack: barcode label
- Control beverage, graphic snack (Experimental): The participant will see fruit drinks with no nutrition claims (task 1). They will see a snack with a graphic label (image of sugar cubes in a cup) along with the text "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Control Drink: No nutrition claim; Behavioral: Experimental snack: Graphic warning
- Claim 1 beverage, text snack (Experimental): The participant will see fruit drinks with the nutrition claim "No Artificial Sweeteners" (task 1). They will see a snack with a text warning "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Experimental snack: Text warning
- Claim 1 beverage, control snack (Experimental): The participant will see fruit drinks with the nutrition claim "No Artificial Sweeteners" (task 1). They will see a snack with a barcode label (control label) (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Control snack: barcode label
- Claim 1 beverage, graphic snack (Experimental): The participant will see fruit drinks with the nutrition claim "No Artificial Sweeteners" (task 1). They will see a snack with a graphic label (image of sugar cubes in a cup) along with the text "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Experimental snack: Graphic warning
- Claim 2 beverage, text snack (Experimental): The participants will see fruit drinks with the nutrition claim "100% Vitamin C daily value" (task 1). They will see a snack with a text warning "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Experimental snack: Text warning
- Claim 2 beverage, control snack (Experimental): The participants will see fruit drinks with the nutrition claim "100% Vitamin C daily value" (task 1). They will see a snack with a barcode label (control label) (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Control snack: barcode label
- Claim 2 beverage, graphic snack (Experimental): The participants will see fruit drinks with the nutrition claim "100% Vitamin C daily value" (task 1). They will see a snack with a graphic label (image of sugar cubes in a cup) along with the text "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Experimental snack: Graphic warning
- Claim 3 beverage, text snack (Experimental): The participants will see fruit drinks with the nutrition claim "100% All Natural" (task 1). They will see a snack with a text warning "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Experimental snack: Text warning
- Claim 3 beverage, control snack (Experimental): The participants will see fruit drinks with the nutrition claim "100% All Natural" (task 1). They will see a snack with a barcode label (control label) (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Control snack: barcode label
- Claim 3 beverage, graphic snack (Experimental): The participants will see fruit drinks with the nutrition claim "100% All Natural" (task 1). They will see a snack with a graphic label (image of sugar cubes in a cup) along with the text "WARNING: High in added sugar" (task 2).
  Interventions: Behavioral: Experimental Drink: Nutrition claim on fruit drinks; Behavioral: Experimental snack: Graphic warning

INTERVENTIONS:
Behavioral: Experimental Drink: Nutrition claim on fruit drinks — Fruit drink contains a nutrition claim (task 1)
  Arms: Claim 1 beverage, control snack; Claim 1 beverage, graphic snack; Claim 1 beverage, text snack; Claim 2 beverage, control snack; Claim 2 beverage, graphic snack; Claim 2 beverage, text snack; Claim 3 beverage, control snack; Claim 3 beverage, graphic snack; Claim 3 beverage, text snack
Behavioral: Control Drink: No nutrition claim — Fruit drinks does not contain a nutrition claim (task 1)
  Arms: Control beverage, control snack; Control beverage, graphic snack; Control beverage, text snack
Behavioral: Experimental snack: Text warning — The snack contains a text warning (task 2)
  Arms: Claim 1 beverage, text snack; Claim 2 beverage, text snack; Claim 3 beverage, text snack; Control beverage, text snack
Behavioral: Experimental snack: Graphic warning — The snack contains a graphic warning (task 2)
  Arms: Claim 1 beverage, graphic snack; Claim 2 beverage, graphic snack; Claim 3 beverage, graphic snack; Control beverage, graphic snack
Behavioral: Control snack: barcode label — The snack contains a neutral barcode label (task 2)
  Arms: Claim 1 beverage, control snack; Claim 2 beverage, control snack; Claim 3 beverage, control snack; Control beverage, control snack

SUMMARY:
Purpose: Examine the impact of nutrition claims on parents' decisions to purchase fruit drinks in a randomized controlled trial in an online virtual convenience store (task 1) and examine the impact of added sugar warnings on parents' snack purchasing decisions in a randomized controlled trial in an online virtual convenience store.

Participants: Participants will consist of approximately 2,500 individuals 18 and older with at least one child ages 1-5. The child 1-5 who had their birthday most recently must have consumed at least one fruit drink in the previous week. Additionally, they will live in the United States and identify as non-Hispanic black, non-Hispanic white, or Hispanic. The panel research company Kantar will recruit individuals from its pool of potential individuals.

Procedures (methods): The investigators will randomize participants to one of 12 versions of a virtual convenience store (iShoppe) and then the participants will complete two shopping tasks in the store. They will select two beverages (task 1) for their child 1-5 who had their birthday most recently, and they will select a snack (task 2) for that same child. After completing the shopping tasks, the participant will complete a survey in Qualtrics. The survey will ask a series of questions about the beverages and snacks (e.g., perceived healthfulness, perceived appeal, intentions to consume products). Questions will also include standard demographic and health related variables.

DETAILED DESCRIPTION:
There are major racial-ethnic disparities in the US childhood obesity epidemic. Among children age 1-5 years, Black children are twice as likely to be obese and Latino children are three times as likely to be obese compared to White children. Sugar-sweetened beverage (SSB) and processed food consumption are major drivers of the childhood obesity epidemic, and an important driver of racial-ethnic obesity disparities. Policies to reduce marketing and require warning labels are important strategies for improving health outcomes among US parents and children at risk for obesity. Understanding the impact of nutrition claims on fruit drink purchases among Black and Latino parents is especially important given pre-existing disparities in early childhood SSB consumption and obesity. However, little is known about the relationship between nutrition claims and SSB purchases among racial-ethnic minorities. Thus, it is important to understand the effect of nutrition claims on racial-ethnic minority parents' purchases of fruit drinks. Another key research gap relates to the impact of warning labels for processed food among this population. Thus, in this study the investigators also aim to test warning labels on food/snack products as part of this study.

Setting: The trial will take place in a virtual convenience store setting created for researchers to examine how store and product characteristics influence consumer purchases in a controlled but realistic environment.

Recruitment: Participants will be recruited online through Kantar's currently available panel participants. Interested potential participants will complete a screener online, and if they are eligible, they will be redirected to the consent form.

Informed consent: Participants will view an online consent form prior to participating in the study, They will acknowledge their consent by proceeding onto the study.

Randomization: After acknowledging consent, participants will be randomized to one of 12 versions of the store(see trial arms). Participants will have an equal chance to be randomized to one of the arms of the store.

Assessment: Participants will enter the virtual convenience store and be given a shopping task to select 2 beverages (task 1) for their child age 1-5 who celebrated their birthday most recently. The participant will have to select between 100% grape juice and a grape-flavored fruit drink, and they will have to select between water and an apple-flavored fruit drink. After selecting two beverages, the participant will then be directed to complete a snack shopping task (task 2). After completing the two shopping tasks, the participant will be redirected to an online survey to complete. Participation in the study will last approximately 15-18 minutes.

Trial arms: All participants will complete two shopping tasks where they have to (1) choose between a grape fruit drink and a 100% grape juice, and choose between an apple fruit drink and water, and (2) choose between a snack with a nutrient warning label or a snack with no warning label. There will be 4 versions of the fruit drinks that participants will be randomized to. They will see either a fruit drink with no claim (control) or a fruit drink with 1 of 3 claims ("No artificial sweeteners," "100% vitamin c daily value," "100% all natural"). For the snack with the nutrient warning label, participants will see either a control label (barcode) or a nutrient warning label (text or graphic).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Currently reside in the US
* Be a Kantar panel member
* have at least one child aged 1-5
* Child 1-5 with the most recent birthday must have consumed at least one fruit drink in the previous week (7 days)
* Self-identify as non-Hispanic white, non-Hispanic black, or Hispanic any race

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2374 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Hall, PhD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Carolina Population Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taillie LS, Higgins ICA, Lazard AJ, Miles DR, Blitstein JL, Hall MG. Do sugar warning labels influence parents' selection of a labeled snack for their children? A randomized trial in a virtual convenience store. Appetite. 2022 Aug 1;175:106059. doi: 10.1016/j.appet.2022.106059. Epub 2022 May 5. PMID 35526703
- [Derived] Hall MG, Lazard AJ, Higgins ICA, Blitstein JL, Duffy EW, Greenthal E, Sorscher S, Taillie LS. Nutrition-related claims lead parents to choose less healthy drinks for young children: a randomized trial in a virtual convenience store. Am J Clin Nutr. 2022 Apr 1;115(4):1144-1154. doi: 10.1093/ajcn/nqac008. PMID 35040866

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Beverage, Text Snack | Control Beverage, Control Snack | Control Beverage, Graphic Snack | Claim 1 Beverage, Text Snack | Claim 1 Beverage, Control Snack | Claim 1 Beverage, Graphic Snack | Claim 2 Beverage, Text Snack | Claim 2 Beverage, Control Snack | Claim 2 Beverage, Graphic Snack | Claim 3 Beverage, Text Snack | Claim 3 Beverage, Control Snack | Claim 3 Beverage, Graphic Snack
Started | 200 | 205 | 199 | 197 | 199 | 195 | 194 | 193 | 214 | 198 | 192 | 188
Completed | 185 | 190 | 190 | 183 | 191 | 180 | 184 | 177 | 195 | 188 | 183 | 173
Not Completed | 15 | 15 | 9 | 14 | 8 | 15 | 10 | 16 | 19 | 10 | 9 | 15

BASELINE CHARACTERISTICS:
Population: Data reported for those participants who completed the entire trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Beverage, Text Snack | Control Beverage, Control Snack | Control Beverage, Graphic Snack | Claim 1 Beverage, Text Snack | Claim 1 Beverage, Control Snack | Claim 1 Beverage, Graphic Snack | Claim 2 Beverage, Text Snack | Claim 2 Beverage, Control Snack | Claim 2 Beverage, Graphic Snack | Claim 3 Beverage, Text Snack | Claim 3 Beverage, Control Snack | Claim 3 Beverage, Graphic Snack | Total
Number analyzed (Participants) | 185 | 190 | 190 | 183 | 191 | 180 | 184 | 177 | 195 | 188 | 183 | 173 | 2219
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
  Age: Between 18 and 65 years | 184 | 190 | 190 | 183 | 190 | 180 | 184 | 177 | 194 | 188 | 181 | 172 | 2213
  Age: >=65 years | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data reported for those who disclosed this information.
  Participants
    Gender: number analyzed (Participants) | 182 | 190 | 188 | 176 | 185 | 177 | 180 | 169 | 191 | 183 | 178 | 172 | 2171
    Gender: Man | 56 | 61 | 67 | 63 | 70 | 69 | 66 | 58 | 62 | 75 | 63 | 58 | 768
    Gender: Woman | 126 | 129 | 121 | 113 | 115 | 108 | 114 | 111 | 128 | 108 | 115 | 114 | 1402
    Gender: Transgender or other gender identity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 63 | 64 | 62 | 56 | 53 | 67 | 62 | 62 | 66 | 58 | 62 | 735
  Not Hispanic or Latino | 125 | 127 | 126 | 121 | 135 | 127 | 117 | 115 | 133 | 122 | 125 | 111 | 1484
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 1 | 1 | 0 | 2 | 15
  Asian | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 5
  Black or African American | 42 | 49 | 41 | 39 | 32 | 39 | 35 | 38 | 46 | 32 | 39 | 40 | 472
  White | 129 | 124 | 137 | 131 | 149 | 128 | 132 | 126 | 136 | 139 | 123 | 117 | 1571
  More than one race | 5 | 5 | 5 | 4 | 2 | 5 | 2 | 3 | 2 | 2 | 7 | 4 | 46
  Unknown or Not Reported | 9 | 9 | 4 | 7 | 6 | 5 | 11 | 7 | 7 | 12 | 10 | 8 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Selected the Grape-Flavored Fruit Drink (Fruit Drink Experimental Task 1)
Description: Measured as percent of participants selecting grape-flavored fruit drink rather than 100% grape juice (objectively measured).
Time Frame: During virtual shopping task which will last ~5 minutes
Measure: Number; unit: percentage of participants
Groups:
- Control Beverage: The participant will see fruit drinks with no nutrition claims (task 1).
  Control Drink: No nutrition claim: Fruit drinks does not contain a nutrition claim (task 1)
- Claim 1 Beverage: The participant will see fruit drinks with the nutrition claim "No Artificial Sweeteners" (task 1).
  Experimental Drink: Nutrition claim on fruit drinks: Fruit drink contains a nutrition claim (task 1)
- Claim 2 Beverage: The participants will see fruit drinks with the nutrition claim "100% Vitamin C daily value" (task 1).
  Experimental Drink: Nutrition claim on fruit drinks: Fruit drink contains a nutrition claim (task 1)
- Claim 3 Beverage: The participants will see fruit drinks with the nutrition claim "100% All Natural" (task 1).
  Experimental Drink: Nutrition claim on fruit drinks: Fruit drink contains a nutrition claim (task 1)
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 565 | 554 | 556 | 544
percentage of participants | 32 | 45 | 51 | 54
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for statistical significance is < 0.05

2. Primary Outcome: Percent of Participants Who Selected the Lower Sugar Granola Snack (Snack Experimental Task 2)
Description: Measured as percent of participants selecting lower sugar granola snack rather than higher sugar granola snack (objectively measured).
Time Frame: During virtual shopping task which will last ~5 minutes
Measure: Number; unit: percentage of participants
Groups:
- Control Snack: The participant will see a snack with a barcode label (control label)
  Control snack: barcode label: The snack contains a neutral barcode label
- Text Snack: The participant will see a snack with a text warning "WARNING: High in added sugar"
  Experimental snack: Text warning: The snack contains a text warning
- Graphic Snack: The participant will see a snack with a graphic label (image of sugar cubes in a cup) along with the text "WARNING: High in added sugar" (task 2).
  Experimental snack: Graphic warning: The snack contains a graphic warning
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 741 | 740 | 738
percentage of participants | 66 | 79 | 82
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; snacks with warning compared to control snack; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for statistical significance is < 0.05

3. Secondary Outcome: Percent of Participants Who Misperceive That the Fruit Drink Does Not Have Added Sugar (Fruit Drink Experimental Task 1)
Description: The percent of participants who hold the misperception that the fruit drink does not have added sugar. Measured by response to the question, "Do you think this beverage has added sugar?" Response options are yes/no. Misperception coded as "no."
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question
Measure: Number; unit: percentage of participants
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 540 | 544 | 536
percentage of participants | 12 | 42 | 22 | 47
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for statistical significance is < 0.05

4. Secondary Outcome: Percent of Participants Who Misperceive That the Fruit Drink is 100% Fruit Juice (Fruit Drink Experimental Task 1)
Description: The percent of participants who hold the misperception that the fruit drink is 100% fruit juice. Measured by response to the question, "Do you think this beverage is 100% fruit juice?" Response options are yes/no. Misperception coded as "yes."
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question
Measure: Number; unit: percentage of participants
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 541 | 544 | 536
percentage of participants | 22 | 36 | 35 | 56
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Logistic — The a priori threshold for statistical significance is < 0.05

5. Secondary Outcome: Number of Teaspoons of Added Sugar Participants Think the Fruit Drink Contains (Fruit Drink Experimental Task 1)
Description: Amount of added sugar people think the product contains. Measured by response to the questions, "A can of regular soda contains 8 teaspoons of added sugar. How many teaspoons of added sugar do you think this beverage has?" Response is free text entry limited to 0-100 (# of teaspoons). This question is only asked if the participant believes the product has added sugar (see outcome 3).
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: This question is only asked of those participants who believe the product has added sugar.
Measure: Mean (Standard Deviation); unit: teaspoons
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 495 | 311 | 427 | 282
teaspoons | 6.4 (3.8) | 5.8 (3.4) | 5.7 (3.8) | 5.9 (4.4)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; Beverages with claim compared to control beverage; Test type: Superiority; p < 0.01, Regression, Linear — The a priori threshold for statistical significance is < 0.05

6. Secondary Outcome: Mean Percent of Fruit Juice That Participants Believe the Fruit Drink Contains (Fruit Drink Experimental Task 1)
Description: The mean percentage of fruit juice participants think the product contains. Measured by response to the question, "What percentage of this beverage do you think is fruit juice?" Response is a sliding scale 0 - 100 (percent fruit juice). This question is only asked if the participant does not believe the drink is 100% fruit juice (see outcome 4).
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: This question is only asked of those participants who believe the product is not 100 percent fruit juice.
Measure: Mean (Standard Deviation); unit: percentage of fruit juice
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 437 | 344 | 355 | 236
percentage of fruit juice | 35.4 (23.0) | 46.3 (24.4) | 40.8 (24.7) | 43.9 (25.4)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

7. Secondary Outcome: Perceived Misleadingness of Fruit Drink (Fruit Drink Experimental Task 1)
Description: Perceived misleadingness of the fruit drink as determined by asking the question, "This beverage is 20% fruit juice and contains 39 grams of added sugar. How misleading do you think the information on this product is?" The response options are on a scale: 1 = Not at all misleading…5 = Extremely misleading.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Claim 3 Beverage: The participants will see fruit drinks with the nutrition claim "100% All Natural" (task 1).
  Experimental Drink: Nutrition claim on fruit drinks: Frui
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 540 | 544 | 536
score on a scale | 3.3 (1.3) | 3.7 (1.3) | 3.7 (1.2) | 3.9 (1.2)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

8. Secondary Outcome: Perceived Product Healthfulness of Fruit Drink for Child's Daily Consumption (Fruit Drink Experimental Task 1)
Description: Perceived product healthfulness as determined by asking the question, "How healthy or unhealthy would it be for [child you shopped for] to drink this beverage every day?" The response options are on a scale: 1 = Very unhealthy...5= Very healthy.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 545 | 547 | 539
score on a scale | 3.3 (1.3) | 3.6 (1.2) | 3.7 (1.2) | 3.8 (1.1)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

9. Secondary Outcome: Interest in Giving the Fruit Drink to One's Child (Fruit Drink Experimental Task 1)
Description: Interest in giving fruit drinks to one's child as determined by asking the question, "How likely would you be to give this beverage to your child?" The response options are on a scale: 1 = Not at all likely…5 = Extremely likely)
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 545 | 547 | 539
score on a scale | 3.4 (1.2) | 3.7 (1.1) | 3.7 (1.2) | 3.8 (1.1)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

10. Secondary Outcome: Percent of Participants Who Selected Apple-flavored Fruit Drink (Fruit Drink Experimental Task 1)
Description: Measured as percent of participants selecting apple-flavored fruit drink rather than water (objectively measured).
Time Frame: During virtual shopping task which will last ~5 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 565 | 554 | 556 | 544
percentage of participants | 55 | 61 | 60 | 62
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.01, Regression, Logistic — The a priori threshold for statistical significance is < 0.05

11. Secondary Outcome: Perceived Appeal of Fruit Drink (Fruit Drink Experimental Task 1)
Description: Perceived appeal of fruit drink as determined by asking the question, "How appealing would your child find this beverage?" The response options are on a scale: 1 = Very unappealing…5=Very appealing.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 545 | 547 | 539
score on a scale | 4.1 (1.0) | 4.2 (0.9) | 4.3 (0.8) | 4.2 (0.9)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.01, Regression, Linear — The a priori threshold for statistical significance is < 0.05

12. Secondary Outcome: Interest in Consuming the Fruit Drink (Fruit Drink Experimental Task 1)
Description: Interest in consuming the fruit drink as determined by asking the questions, "How likely would you be to drink. this beverage?" The response options are on a scale: 1 = Not at all likely…5= Extremely likely.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 545 | 546 | 539
score on a scale | 3.3 (1.4) | 3.5 (1.3) | 3.5 (1.3) | 3.6 (1.3)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

13. Secondary Outcome: Relative Harm of the Fruit Drink Compared to Soda (Fruit Drink Experimental Task 1)
Description: Relative harm of the fruit drink compared to soda as determined by asking the question, "Compared to regular (non-diet) soda, this beverage is…" The response options are on a scale: 1 = Much less healthy…5 = Much healthier.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 540 | 544 | 536
score on a scale | 3.6 (0.9) | 3.9 (0.8) | 3.9 (0.9) | 4.0 (0.9)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

14. Secondary Outcome: Relative Harm of the Fruit Drink Compared to 100% Fruit Juice (Fruit Drink Experimental Task 1)
Description: Relative harm of the fruit drink compared to 100% fruit juice as determined by asking the question, "Compared to 100% fruit juice, this beverage is…" The response options are on a scale: 1 = Much less healthy…5 = Much healthier.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Beverage | Claim 1 Beverage | Claim 2 Beverage | Claim 3 Beverage
Number analyzed (Participants) | 561 | 540 | 544 | 536
score on a scale | 2.3 (1.3) | 2.8 (1.2) | 2.8 (1.4) | 3.2 (1.3)
Statistical Analysis 1: Comparison: Control Beverage vs Claim 1 Beverage vs Claim 2 Beverage vs Claim 3 Beverage; beverages with claim compared to control beverage; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

15. Secondary Outcome: Perceived Product Healthfulness of Snack (Snack Experimental Task 2)
Description: Perceived product healthfulness of the snack as determined by asking, "How healthy would it be for your child to eat this snack every day?" The response options are on a scale: 1=very unhealthy…5=very healthy.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 730 | 728 | 728
score on a scale | 3.9 (0.9) | 2.6 (1.5) | 2.5 (1.4)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

16. Secondary Outcome: Product Appeal of Snack for One's Child (Snack Experimental Task 2)
Description: Product appeal of the snack as determined by asking, "How appealing would your child find this snack?" The response options are on a scale: 1=very unappealing…5=very appealing.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 730 | 727 | 727
score on a scale | 3.7 (1.1) | 3.5 (1.3) | 3.5 (1.3)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

17. Secondary Outcome: Participant Intentions to Give Snack to One's Child (Snack Experimental Task 2)
Description: Intentions to give snack to child as determined by asking, "How likely would you be to give this snack to your child?" The response options are on a scale: 1=not at all likely…5=extremely likely.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 729 | 727 | 728
score on a scale | 3.6 (1.1) | 2.6 (1.4) | 2.5 (1.4)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

18. Secondary Outcome: Intentions to Purchase the Snack (Snack Experimental Task 2)
Description: Intentions to purchase snack as determined by asking, "How likely would you be to buy this snack in the next week?" The response options are on a scale: 1=not at all likely…5=extremely likely.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 730 | 727 | 729
score on a scale | 3.4 (1.2) | 2.5 (1.4) | 2.4 (1.4)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

19. Secondary Outcome: Intentions to Consume the Snack (Snack Experimental Task 2)
Description: Intentions to consume snack as determined by asking, "How likely would you be to consume this snack?" The response options are on a scale: 1=not at all likely….5=extremely likely.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 730 | 728 | 727
score on a scale | 3.5 (1.2) | 2.7 (1.4) | 2.6 (1.4)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

20. Secondary Outcome: Percent of Participants Able to Identify the Healthier Snack (Snack Experimental Task 2)
Description: Correct identification of healthier snack, as measured by response to the question "Which of these snacks would be healthier for your child?" Response options include the snack product with the added sugar warning and the snack product without the sugar warning.
  snack without the added sugar warning = healthier snack
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question
Measure: Number; unit: percentage of participants
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 726 | 725 | 726
percentage of participants | 59 | 87 | 87
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

21. Secondary Outcome: Percent of Participants Able to Identify the Snack With Higher Amount of Added Sugar (Snack Experimental Task 2)
Description: Correct identification of snack with higher added sugar, as measured by response to the question "Which of these snacks is higher in added sugar?" Response options include the snack product with the added sugar warning and the snack product without the sugar warning.
  snack with added sugar warning = snack with higher amount of added sugar
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question
Measure: Number; unit: percentage of participants
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 726 | 726 | 728
percentage of participants | 44 | 79 | 74
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

22. Secondary Outcome: Percent of Participants Who Intend to Purchase the Snack With Higher Added Sugar (Snack Experimental Task 2)
Description: Intentions to purchase snack with higher added sugar, as measured by response to the question, "Which of these snacks would you most want to buy for your child?" Response options include the snack product with the added sugar warning and the snack product without the sugar warning.
  snack with added sugar warning = snack with higher amount of added sugar
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question
Measure: Number; unit: percentage of participants
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 726 | 727 | 727
percentage of participants | 38 | 12 | 13
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

23. Secondary Outcome: Perceived Message Effectiveness of Snack (Snack Experimental Task 2)
Description: Perceived message effectiveness as measured by average response to three questions:
  1. How much does this label make you concerned about the health effects of consuming this product? The response options are on a scale: 1=not at all…5=a great deal.
  2. How much does this label make consuming this product seem unpleasant to you? The response options are on a scale: 1=not at all…5=a great deal.
  3. How much does this label discourage you from wanting to consume this product? The response options are on a scale: 1=not at all…5=a great deal.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Graphic Snack: The participant will see a snack with a graphic label (image of sugar cubes in a cup) along with the text "WARNING: High in added sugar" Experimental snack: Graphic warning: The snack contains a graphic warning
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 729 | 724 | 728
score on a scale | 2.3 (1.3) | 4.2 (0.9) | 4.3 (0.8)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

24. Secondary Outcome: Social Reactions to Snack (Snack Experimental Task 2)
Description: Anticipated social reactions as measured by response to questions, "How likely are you to talk about this label with others in the next week?" The response options are on a scale: 1= not at all likely…5=extremely likely.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 730 | 727 | 729
score on a scale | 2.2 (1.4) | 3.1 (1.4) | 3.1 (1.4)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

25. Secondary Outcome: Percent of Participants Who Learned Something New About the Snack (Snack Experimental Task 2)
Description: Percent who learned something new about the snack as measured by the question, "Did you learn something new from this label" The response options are yes/no. Yes indicates the participant learned something new.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Number; unit: percentage of participants
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 728 | 727 | 728
percentage of participants | 24 | 75 | 77
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

26. Secondary Outcome: Snack Grabbed the Participant's Attention (Snack Experimental Task 2)
Description: The extent to which the snack grabbed the participant's attention as measured by the question, "How much does this label grab your attention?" The response options are on a scale:1=not at all…5=a great deal.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 728 | 727 | 729
score on a scale | 2.5 (1.4) | 4.4 (0.9) | 4.4 (0.9)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

27. Secondary Outcome: Label on Snack Makes Participant Feel Scared (Snack Experimental Task 2)
Description: The extent to which the snack made the participant feel scared as measured by the questions, "How much does this label make you feel scared?" The response options are on a scale: 1=not at all…5=a great deal.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 728 | 726 | 728
score on a scale | 1.9 (1.3) | 3.3 (1.3) | 3.4 (1.3)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

28. Secondary Outcome: Thinking About the Health Effects of the Snack (Snack Experimental Task 2)
Description: The extent to which the snack made the participant think about the health effects of the snack as measured by the question, "How much does this label make you think about the health problems caused by eating this snack?" The response options are on a scale: 1=not at all…5=a great deal.
Time Frame: 13-15 minutes post-test computer survey following the ~5 minute virtual shopping task.
Population: Data provided for those participants who responded to this optional question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Snack | Text Snack | Graphic Snack
Number analyzed (Participants) | 728 | 727 | 729
score on a scale | 2.1 (1.4) | 4.1 (1.0) | 4.1 (1.0)
Statistical Analysis 1: Comparison: Control Snack vs Text Snack vs Graphic Snack; warning snacks compared to control snack; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is < 0.05

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed Consent through study completion, an approximate total of up to 20 minutes.
Arm/Group | Control Beverage, Text Snack | Control Beverage, Control Snack | Control Beverage, Graphic Snack | Claim 1 Beverage, Text Snack | Claim 1 Beverage, Control Snack | Claim 1 Beverage, Graphic Snack | Claim 2 Beverage, Text Snack | Claim 2 Beverage, Control Snack | Claim 2 Beverage, Graphic Snack | Claim 3 Beverage, Text Snack | Claim 3 Beverage, Control Snack | Claim 3 Beverage, Graphic Snack
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/205 | 0/199 | 0/197 | 0/199 | 0/195 | 0/194 | 0/193 | 0/214 | 0/198 | 0/192 | 0/188
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/205 | 0/199 | 0/197 | 0/199 | 0/195 | 0/194 | 0/193 | 0/214 | 0/198 | 0/192 | 0/188
Other Adverse Events (participants affected / at risk) | 0/200 | 0/205 | 0/199 | 0/197 | 0/199 | 0/195 | 0/194 | 0/193 | 0/214 | 0/198 | 0/192 | 0/188

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04381481/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04381481/SAP_000.pdf